CLINICAL TRIAL: NCT05858177
Title: The Efficacy and Safety of Temozolomide in Patients With Metastatic Pheochromocytoma or Paraganglioma
Brief Title: The Efficacy and Safety of Temozolomide in Patients With MPPGL
Acronym: MPPGL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06086-03
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: Pheochromocytoma, Metastatic; Paraganglioma, Malignant; Pheochromocytoma Malignant
Keywords: Pheochromocytoma or Paraganglioma; metastasis; Temozolomide
MeSH Terms: conditions — Pheochromocytoma; Neoplasm Metastasis; Paraganglioma, Extra-Adrenal; Paraganglioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temozolomide (Other): TMZ was given orally per day for 5 days, every 28 days until disease progression or intolerable toxicities.
  Interventions: Drug: Temozolomide capsule

INTERVENTIONS:
Drug: Temozolomide capsule — Temozolomide was given orally per day for 5 days, every 28 days until disease progression or intolerable toxicities.
  Other Names: Temozolomide

SUMMARY:
Metastatic pheochromocytoma / paraganglioma (MPP) are rare while the prognosis was poor. Temozolomide (TMZ) is a novel oral alkylation chemotherapeutic agent. TMZ has been recommended in National Comprehensive Cancer Network (NCCN) Guidelines Version 1.2019 for treating MPP patients.However, studies investigating TMZ efficacy in MPP patients are extremely limited. The largest study involved only 15 patients till date. The safety and efficacy of TMZ treatment in MPP patients need to be verified in larger studies.

DETAILED DESCRIPTION:
Patients with histologically or radiologically confirmed MPP were enrolled. TMZ was administered orally at an initial daily dose of 150 mg/m2 per day for 5 days, every 28 days. In patients with a good tolerance during the first cycle, the dose was increased to 200 mg/m2 per day for 5 days, every 28 days. Plasma normetanephrine and metanephrine (MNs), 24-hour urinary catecholamine excretion (24hCA) and neuron specific enolase (NSE) were measured at baseline and every 1-3 cycle. Contrast-enhanced computed tomography（CT ）of chest, abdomen and pelvis were used to assess measurable target lesions at baseline and every 3 cycles. For patients who only had bone metastases or no measurable target lesions, TMZ efficacy was evaluated by 18F-fluorodeoxyglucose (18F-FDG-PET/CT). The primary endpoint was objective response rate (ORR) per Response Evaluation Criteria In Solid Tumors（RECIST) 1.1/PERCIST1.0. Secondary endpoints included biochemical (catecholamine levels) response rate (BRR), progression-free survival (PFS) and safety. The investigators will try to explore which patients are more suitable for TMZ treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with metastatic pheochromocytomas and paragangliomas. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

Estimated life expectancy longer than 6 months. Having normal organ function as defined by hemoglobin levels ≥10 g/dL, absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 80 x 109/L, total bilirubin ≤1.5 institutional upper limit, aspartate aminotransferase ≤5 institutional upper limit, alanine aminotransferase ≤5 institutional upper limit, and serum creatinine <3.0 mg/dL.

Exclusion Criteria:

Didn't meet eligibility for organ function. Pregnancy or breastfeeding. Uncontrolled congestive heart failure and severe infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
disease control rate (DCR) | At the end of Cycle 3 (each cycle is 28 days)
  Defined for all patients whose tumor met the criteria of CR or PR or stable disease(SD)
objective response rate (ORR) | At the end of Cycle 3 (each cycle is 28 days)
  Defined for all patients whose tumor met the criteria of Complete Response (CR)and Partial Response (PR)

SECONDARY OUTCOMES:
progression-free survival (PFS) | At least 1 cycle(each cycle is 28 days), up to 100 weeks,From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS is defined as the time from the first day of treatment to the first documented disease progression per RECIST 1.1 criteria and the Kaplan-Meier curve. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.
biochemical response | At the end of Cycle 1 (each cycle is 28 days)
  An effective response of 24hCA, MNs or NSE meant that the concentration decreased by more than 40% than the baseline value or decreased to the normal range
Incidence of adverse events | At the end of Cycle 1 (each cycle is 28 days)
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Anli Tong, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No